CLINICAL TRIAL: NCT01597843
Title: Working With Veterans Organizations to Encourage Use of My HealtheVet
Brief Title: Veterans Service Organizations and My HealtheVet (MHV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: The American Legion Department of Wisconsin (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RRP 11-408
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension; Hyperlipidemia; Coronary Artery Disease; Diabetes Mellitus
Keywords: education; self care; peer group; Computers; Attitude to computers
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Coronary Artery Disease; Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- First educational intervention group (Experimental): Group that receives intervention first. The intervention is a series of training sessions, in person and on line, to educate post superusers who will in turn educate post members on the utility and mechanics of use of MHV.
  Interventions: Other: Education
- Second intervention group (Experimental): This arm receives a series of training sessions over study months 6-9. The training sessions are in person and on line and are directed at post superusers who will in turn educate post members on the utility and mechanics of use of MHV. They complete survey rounds 1 and 2 before the training and survey round 3 after the training.
  Interventions: Other: Education
- Education after data collection complete (No Intervention): This group received a similar intervention, but after all quantitative data collection complete.

INTERVENTIONS:
Other: Education — Series of training sessions, in person and on line, to educate post superusers who will in turn educate post members on the utility and mechanics of use of MHV.
  Other Names: Post education
  Arms: First educational intervention group; Second intervention group

SUMMARY:
This project will design, deliver, and evaluate a peer support intervention that will help veterans become familiar with and register for Veterans Health Administration (VHA) My HealtheVet (MHV). It will lay the groundwork for 2 types of future projects. First, the investigators will develop materials that can be used in other settings to increase registration, authentication, and meaningful use of MHV. Second, it will allow us to develop and study interventions that use informed, peer-supported Internet use to improve health behaviors and outcomes among veterans.

DETAILED DESCRIPTION:
BACKGROUND/RATIONALE: Despite the promise of electronic health resources, there is evidence that they have not led to the improved self management that many envisioned. There is evidence for this from a variety of sources, including the Veterans Health Administration (VHA). Although there is appropriate attention to improving the functionality and ease of use of the system, a key barrier is patient acceptance and familiarity. Peer support, particularly in group settings, can improve health-related behaviors. Such approaches may increase and improve MHV use.

OBJECTIVES: Our goal in the present project is to develop and test a peer-based mechanism to increase MHV use by member of veterans service organizations (VSO) such as the American Legion. The investigators will address 3 specific aims:

1. To demonstrate that trained members of VSO can provide basic MHV education and support within their VSO unit using mobile computers.
2. To demonstrate that this intervention increases MHV registration, in person authentication (IPA), and reported use of MHV among veteran post members.
3. To create clear, concise, and portable resources that will make it possible to replicate this process in other VSO units or other community settings.

METHODS: This implementation study is a quasi-randomized intervention with delayed controls. Working with the leadership of selected veterans groups, the investigators will identify 12 posts that have the appropriate resources and interests to serve as pilot posts for the present project. The investigators will train 2 peer mentors (super-users or SU) from 4 of these posts using adaptations of the peer training approach the investigators used for a previous project. The investigators will work with the SU to install computers with wireless broadband Internet access at their posts. The investigators will load the computers with software that documents unique sessions, sites visited, and amount of time at each site. The investigators will help the SU provide lessons regarding MHV use to his/her fellow post members at 4 monthly post meetings. After 4 months, the investigators will move the computers to the next 4 posts and repeat the intervention. Finally, the investigators will move the computers to the last 4 posts, providing remote support and our training materials to the SU at those posts. The investigators will use computer tracking data, surveys, focus groups, and interviews to assess the impact of the program. The investigators will test changes in registration, IPA, and use with before and after surveys. Our analysis will adjust for clustering within posts. The investigators will transcribe our focus groups and interviews verbatim and analyze them using a case study approach.

ELIGIBILITY:
Inclusion Criteria:

Two steps, first a post is enrolled, then a member participates.

Post eligible if:

* The post leadership agrees that the post will support participation.
* Two or more members of the post agree to serve as MHV super-users.
* There is an identifiable location within the post for the computer.

Member eligible if:

* Member of post
* Attends the meeting at which the survey is administered

Exclusion Criteria:

* Does not consent to survey
* Does not attend meeting where survey administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Whittle, MD MPH, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI
Locations (1):
- Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin, United States

REFERENCES:
- See also: American Legion Website for Department of Wisconsin — http://www.wilegion.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 12 posts at the outset of the study, with the help of the Legion's state leadership. We invited all post members to complete surveys at times 0, 5 months and 10 months. The surveys were distributed by post leadership at a post meeting. We did not obtain informed consent; we obtained no personal identifiers but we obtained post.
Groups:
- Education in First Round: Four of twelve posts were in this group and were randomized to receive a series of training sessions. The training sessions were in person and on line, to educate post superusers who will in turn educate post members on the utility and mechanics of use of MHV. The participants at these 4 posts received the intervention in study months 1-5. They completed survey round 1 before receiving the intervention and survey rounds 2 and 3 after receiving the intervention. The number of participants at any post who showed up to respond to any of the three survey rounds varied.
- Control First Round; Education in Second Round: Four of twelve posts were in this group and were randomized to receive a series of training sessions. The training sessions were in person and on line, to educate post superusers who will in turn educate post members on the utility and mechanics of use of MHV. The participants at these 4 posts received the intervention in study months 6-9. They completed survey rounds 1 and 2 before receiving the intervention and survey round 3 after they received the intervention. The number of participants at any post who showed up to respond to any of the three survey rounds varied.
- Control First Round; Control Second Round; Intervention: Four of twelve posts were in this group and were randomized to receive a series of training sessions. The training sessions were in person and on line, to educate post superusers who will in turn educate post members on the utility and mechanics of use of MHV. The participants at these 4 posts received the intervention in study months 10 - 14. They completed all three survey rounds before receiving the intervention. The number of participants at any post who showed up to respond to any of the three survey rounds varied.
Period: Overall Study
Arm/Group | Education in First Round | Control First Round; Education in Second Round | Control First Round; Control Second Round; Intervention
Started | 79 | 122 | 81
Survey 1 Responses | 45 | 71 | 59
Survey 2 Responses | 52 | 42 | 58
Survey 3 Responses | 65 | 56 | 76
Completed | 79 | 122 | 81
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We included the mean number of post members across the three data collection times as our best measure of participants
Groups:
- Second Intervention Group: The group that receives the intervention second. The intervention is the same as for the first group.
  Education: Series of training sessions, in person and on line, to educate post superusers who will in turn educate post members on the utility and mechanics of use of MHV.
- Total: Total of all reporting groups
Arm/Group | First Educational Intervention Group | Second Intervention Group | Education After Data Collection Complete | Total
Number analyzed (Participants) | 79 | 122 | 81 | 282
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age from self reported survey. We combined data from all three survey rounds to obtain the most stable estimate of age. Note that we do not have data on all people in intervention groups, just the respondents. The mean age presented is at the person level. Thus, for each group, data from all survey respondents in the 4 posts in that group are included.
  Years | 69.9 (10.3) | 65.0 (10.7) | 66.6 (12.4) | 67.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Since the vast majority (> 95%)of members are male, we did not gather gender data. We report them as 100% male, knowing this is likely incorrect.
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 79 | 122 | 81 | 282
Proportion at Educational level [Mean (Standard Deviation); unit: Proportion of participants] — Self report on survey. The mean presented is the mean proportion of all survey responses from each of the posts in each group. We treated all surveys as independent. Thus, the proportion of responses in each category (i.e., Less than high school; High school or GED; college or technical degree; Missing) adds up to 1.0 for each group.
  Proportion of participants
    Less than high school | 0.068 (0.25) | 0.030 (0.17) | 0.057 (0.23) | 0.052 (0.22)
    High school or GED | 0.617 (0.48) | 0.438 (0.50) | 0.674 (0.469) | 0.580 (0.494)
    College or technical degree | 0.241 (0.428) | 0.479 (0.500) | 0.233 (0.423) | 0.315 (0.465)
    Missing | 0.074 (0.262) | 0.053 (0.224) | 0.036 (0.186) | 0.053 (0.224)

OUTCOME MEASURES:

1. Primary Outcome: Registration for MHV
Description: Measured by response to question: Have you ever used My HealtheVet online?
Time Frame: Baseline; After Group 1 Intervention; After Group 2 Intervention
Population: Respondents to first round survey
Measure: Number; unit: Percentage of respondents who use MHV
Groups:
- Education in First Round: Series of training sessions, in person and on line, to educate post superusers who will in turn educate post members on the utility and mechanics of use of MHV. This group received the intervention during study months 1-5, following survey 1, prior to survey rounds 2 and 3.
- Control First Round; Education in Second Round: The intervention was delivered to 3 groups of 4 posts in sequence. The posts in this second round received the intervention over the second study period, from month 6 through month 9. they completed survey rounds 1 and 2 before receiving the intervention, survey round 3 after.
- Control First Round; Control Second Round; Intervention: This group received the intervention in study months 10 - 14. They completed all three survey rounds before receiving the intervention.
Arm/Group | Education in First Round | Control First Round; Education in Second Round | Control First Round; Control Second Round; Intervention
Number analyzed (Participants) | 79 | 122 | 81
Percentage of respondents who use MHV
  Baseline survey | 6.7 | 12.7 | 11.9
  Post first round survey | 25.0 | 7.1 | 12.1
  Post second round survey | 33.9 | 25.0 | 13.2

ADVERSE EVENTS:
Time Frame: Adverse events were not collected as a part of this study
Description: Adverse events were not collected as a part of this study
Arm/Group | Education in First Round | Control First Round; Education in Second Round | Control First Round; Control Second Round; Intervention
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Response rates on surveys were lower than expected. One of the first round intervention posts almost certainly did not deliver anything resembling the planned educational intervention at any point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes